CLINICAL TRIAL: NCT01778322
Title: WEB Clinical Assessment of IntraSaccular Aneurysm Therapy
Acronym: WEBCAST
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP 11-001
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2022-08

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Index Embolization Cohort: WEB Aneurysm Embolization System
  Interventions: Procedure: Intracranial aneurysm embolization

INTERVENTIONS:
Procedure: Intracranial aneurysm embolization — Treatment of intracranial aneurysms

SUMMARY:
The objective of this clinical study is to evaluate clinical utility of the WEB Aneurysm Embolization System used to embolize intracranial aneurysms

DETAILED DESCRIPTION:
The following parameters will be evaluated as part of this study:

* Aneurysm morphology
* Aneurysm size
* For ruptured aneurysms: Hunt and Hess Classification of Subarachnoid Hemorrhage (SAH)
* Size of the embolization device(s) used in the procedure
* Intra-procedural assessment of aneurysm occlusion and flow stasis
* Degree of aneurysm occlusion post-procedure (percentage occlusion, Raymond Scale and other scores as appropriate)
* Aneurysm occlusion durability
* Recanalization rate
* Device-related changes in Modified Rankin Scale from baseline
* Complications/adverse events
* Rebleed/new bleed

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must sign and date an IRB/EC-approved written informed consent prior to initiation of any study procedures

Exclusion Criteria:

* Must not have clinical or angiographic evidence of vasospasm
* Must not have lesion with characteristics unsuitable for endovascular treatment
* Must not have neurologic or psychiatric conditions, which preclude ability to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule
* Must not be concurrently involved in another investigational or post-market study
* Must not have received any investigational device for treatment of the target intracranial aneurysm prior to entry into this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with:
  - Diameter and width of the aneurysm is appropriate size for treatment with the WEB Aneurysm Embolization System per device Instructions for Use
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Durability of occlusion | 6 months
  Evaluated by the Corelab

SECONDARY OUTCOMES:
Recurrence/recanalization rate | 6 months
  Evaluated by the Corelab, based on Raymond Roy occlusion scale
Modified Raymond Scale | 6 months
  Evaluation of patient's functional level of activity by the physician
Percentage occlusion of target aneurysm | 6 months
  Evaluated by the Corelab

OTHER OUTCOMES:
Fluoroscopy time | procedure
  Duration of fluoroscopy time will be recorded during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pierot, MD, Principal Investigator — CHU REIMS
Locations (12):
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Hôpital Beaujon, Clichy
  - CHU Gui de Chauliac, Montpellier
  - CHU Reims Maison Blanche, Reims
  - CHU Purpan, Toulouse
  - CHU Bretonneau, Tours
- Germany (5):
  - Uniklinik Koeln, Cologne
  - Helios Klinikum, Erfurt
  - Klinikum der Johann Wolfgang Goethe Universität, Frankfurt
  - Klinikum Vest GmbH, Recklinghausen
  - Klinikum Stuttgart- Katharinenhospital, Stuttgart
- National Institute of Neurosciences, Budapest, Hungary

REFERENCES:
- [Derived] Pierot L, Szikora I, Barreau X, Holtmannspoetter M, Spelle L, Klisch J, Herbreteau D, Costalat V, Fiehler J, Januel AC, Liebig T, Stockx L, Weber W, Berkefeld J, Moret J, Molyneux A, Byrne J. Aneurysm treatment with the Woven EndoBridge (WEB) device in the combined population of two prospective, multicenter series: 5-year follow-up. J Neurointerv Surg. 2023 Jun;15(6):552-557. doi: 10.1136/neurintsurg-2021-018414. Epub 2022 Jul 8. PMID 35803731
- [Derived] Pierot L, Szikora I, Barreau X, Holtmannspoetter M, Spelle L, Herbreteau D, Fiehler J, Costalat V, Klisch J, Januel AC, Weber W, Liebig T, Stockx L, Berkefeld J, Moret J, Molyneux A, Byrne J. Aneurysm treatment with WEB in the cumulative population of two prospective, multicenter series: 3-year follow-up. J Neurointerv Surg. 2021 Apr;13(4):363-368. doi: 10.1136/neurintsurg-2020-016151. Epub 2020 Jun 12. PMID 32532858
- [Derived] Pierot L, Moret J, Barreau X, Szikora I, Herbreteau D, Turjman F, Holtmannspotter M, Januel AC, Costalat V, Fiehler J, Klisch J, Gauvrit JY, Weber W, Desal H, Velasco S, Liebig T, Stockx L, Berkefeld J, Molyneux A, Byrne J, Spelle L. Safety and efficacy of aneurysm treatment with WEB in the cumulative population of three prospective, multicenter series. J Neurointerv Surg. 2018 Jun;10(6):553-559. doi: 10.1136/neurintsurg-2017-013448. Epub 2017 Sep 30. PMID 28965106
- [Derived] Pierot L, Spelle L, Molyneux A, Byrne J; WEBCAST and French Observatory Investigators. Clinical and Anatomical Follow-up in Patients With Aneurysms Treated With the WEB Device: 1-Year Follow-up Report in the Cumulated Population of 2 Prospective, Multicenter Series (WEBCAST and French Observatory). Neurosurgery. 2016 Jan;78(1):133-41. doi: 10.1227/NEU.0000000000001106. PMID 26552042
- See also: Clinical and Anatomical Follow-up in Patients With Aneurysms Treated With the WEB Device: 1-Year Follow-up Report in the Cumulated Population of 2 Prospective, Multicenter Series (WEBCAST and French Observatory). — http://www.ncbi.nlm.nih.gov/pubmed/26552042
- See also: Safety and efficacy of aneurysm treatment with WEB: results of the WEBCAST study. — http://www.ncbi.nlm.nih.gov/pubmed/26381253
- See also: Aneurysm Treatment With Woven EndoBridge in the Cumulative Population of Three Prospective, Multicenter Series: 2-Year Follow-up — http://www.ncbi.nlm.nih.gov/pubmed/31960052
- See also: Aneurysm treatment with WEB in the cumulative population of two prospective, multicenter series: 3-year follow-up — https://pubmed.ncbi.nlm.nih.gov/32532858/
- See also: Aneurysm treatment with the Woven EndoBridge (WEB) device in the combined population of two prospective, multicenter series: 5-year follow-up — https://jnis.bmj.com/content/early/2022/07/07/neurintsurg-2021-018414
- See also: Safety and Efficacy of Aneurysm Treatment with the WEB: Results of the WEBCAST 2 Study — http://www.ajnr.org/content/38/6/1151